CLINICAL TRIAL: NCT05236205
Title: Antimicrobial Photodynamic Therapy as an Adjunct for Management of Deep Caries Lesions - Study Protocol for a Randomized, Controlled Clinical Trial
Brief Title: Antimicrobial Photodynamic Therapy as an Adjunct for Management of Deep Caries Lesions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UrucumCaries
Record Dates: First submitted 2022-01-21; First posted 2022-02-11 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The clinical evaluations of the carious tissue removal, as well as the microbiological and radiographic analyses, will be performed by examiners blinded to the treatments performed on each tooth.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Experimental): This group will receive the treatment of caries removal with a lowspeed drill (conventional treatment).
  Interventions: Procedure: Caries removal with a lowspeed drill
- Papacarie (Experimental): In this group, partial caries removal with Papacarie will be performed.
  Interventions: Procedure: Partial removal of carious tissue with the administration of Papacarie™
- Papacarie and Bixa orellana extract (Experimental): In this group, partial caries removal with Papacarie and the application of Bixa orellana extract (20%) will be performed.
  Interventions: Procedure: Partial removal of carious tissue with the administration of Papacarie™ and application of Bixa Orellana extract (20%)
- Partial removal with aPDT (Experimental): In this group, partial removal of the carious tissue will be performed, with Papacarie and the application of Bixa orellana extract (20%) with blue LED (aPDT).
  Interventions: Procedure: Partial removal of carious tissue with the administration of Papacarie™, application of Bixa Orellana extract (20%) and LED (aPDT)

INTERVENTIONS:
Procedure: Caries removal with a lowspeed drill — 1. Initial periapical and interproximal radiographs;
  2. Prophylaxis with toothbrush and fluoride toothpaste;
  3. Relative isolation with lip bumper, cotton roll, and aspirator;
  4. Microbiological sampling with ear curette for standardization of volume of carious tissue;
  5. Removal of carious dentin with carbide burs and manual instruments;
  6. Additional microbiological sampling;
  7. Clinical inspection of texture of remaining dentin with an exploratory probe;
  8. Restoration with glass ionomer cement (Ketac Molar Easy Mix - 3M ESPE);
  9. Clinical and radiographic follow-up immediately, 1 week, 1, 3, 6, and 12 months.
  Arms: Control Group
Procedure: Partial removal of carious tissue with the administration of Papacarie™ — 1. Initial radiographs;
  2. Relative isolation;
  3. Microbiological sample with otoscope curette to standardize volume of carious tissue;
  4. Application of Papacarie™ for 5 m inutes, removal of carious tissue around lateral walls of the cavity with noncutting curette and no removal of carious tissue on pulp floor;
  5. Second microbiological sample of remaining dentin with curette;
  6. Clinical evaluation by inspection of texture of remaining dentin with exploratory probe;
  7. Restoration with glass ionomer cement;
  8. Clinical and radiographic follow-up immediately, 1 week, 1, 3, 6, and 12 months after treatment.
  Arms: Papacarie
Procedure: Partial removal of carious tissue with the administration of Papacarie™ and application of Bixa Orellana extract (20%) — 1. Initial radiographs;
  2. Relative isolation;
  3. Microbiological sample with otoscope curette to standardize volume of carious tissue;
  4. Application of Papacarie™ with Bixa Orellana extract (20%) for 5 minutes, removal of carious tissue around lateral walls of the cavity with noncutting curette;
  5. Irradiation of dental tissue for 1 minute on a single point;
  6. Second microbiological sample of remaining dentin with curette;
  7. Clinical evaluation by inspection of texture of remaining dentin with exploratory probe;
  8. Restoration with glass ionomer cement;
  9. Clinical and radiographic follow-up immediately, 1 week, 1, 3, 6, and 12 months after treatment.
  Arms: Papacarie and Bixa orellana extract
Procedure: Partial removal of carious tissue with the administration of Papacarie™, application of Bixa Orellana extract (20%) and LED (aPDT) — 1. Initial radiographs;
  2. Relative isolation;
  3. Microbiological sample with otoscope curette to standardize volume of carious tissue;
  4. Application of Papacarie™ with Bixa Orellana extract (20%) for 5 minutes and the blue light-emitting diode (LED) irradiation with 440-480 nm. Removal of carious tissue around lateral walls of the cavity with noncutting curette;
  5. Irradiation of dental tissue for 1 minute on a single point;
  6. Second microbiological sample of remaining dentin with curette;
  7. Clinical evaluation by inspection of texture of remaining dentin with exploratory probe;
  8. Restoration with glass ionomer cement (Ketac Molar EasyMIx 3M ESPE);
  9. Clinical and radiographic follow-up immediately, 1 week, 1, 3, 6, and 12 months after treatment.
  Arms: Partial removal with aPDT

SUMMARY:
Alternatively to conventional treatments, chemo-mechanical caries removal agents can be used. A modality of treatment that has been increasing in dentistry is antimicrobial photodynamic therapy (aPDT). Bixa orellana, is being researched for application in aPDT. This protocol aims to determine the effectiveness of aPDT with Bixa orellana extract in deep caries lesions. Methods and analysis: A total of 160 teeth with deep occlusal dental caries will be selected and divided in 3 groups: G1 - control group (Caries removal with a lowspeed drill); G2 - Partial Caries Removal with Papacarie; G3 - Partial Caries Removal with Papacarie and application Bixa orellana extract (20%); G4 - Partial Caries Removal with Papacarie and application Bixa orellana extract (20%) with LED (aPDT). After treatment, all the teeth will be restored with glass ionomer cement and followed up clinically and radiographically, with evaluations at immediately, 1 week, 1, 3, 6, and 12 months. Dentin samples before and after treatment will be analyzed microbiologically. The data will be submitted to descriptive statistical analysis of the association between the categorical variables using the chi-square test and Fisher exact text. The Student t test and analysis of variance will be used for the comparison of mean signs and symptoms of reversible pulpitis. Pearson correlation coefficients will be calculated for the analysis of correlations among the continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* Adequate health with no systemic conditions;
* Adequate cooperation;
* Clinically presenting at least 1 permanent molar with an acute, active caries on the dentin not surpassing 2/3 and only involving the occlusal face, with direct view and access as well as no clinical or radiographic signs of pulp involvement.

Exclusion Criteria:

* Systemic adverse health condition;
* Uncooperative behavior;
* Class II, III, IV, or V carious lesion based on Black classification;
* Clinically: caries involving enamel, deficient restorations, small carious lesions on dentin with no access for manual scalers, hidden caries, sign or symptom of pulp involvement, clinical impossibility of restoration;
* Radiographically: evidence of pulp involvement, carious lesion extending beyond 2/3 of dentin.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in Microbiological Evaluation | Baseline and immediately after treatment.
  A sample of caries-affected dentin will be taken from each selected tooth before the removal of the carious tissue. All procedures will be performed in duplicate, and the mean of the counts will be calculated. The results will be expressed in CFU of SM and LB as well as in proportion of streptococcus (% S/VM), SM group (% SM/VM and lactobacilli (% LB/VM) in relation to the total of VM. Immediately after the removal of the carious tissue, samples of the remaining dentin will be taken with a Meyhoefer auricular n° 2 curette and the procedures will be repeated.

SECONDARY OUTCOMES:
Changes in Radiographic evaluation | Baseline, immediately after treatment, 1 week, 1, 3, 6, and 12 months after treatment.
  Periapical and interproximal radiographs will be taken initially and immediately after the procedure. Subsequently, follow up will be performed at immediately, 1 week, 1, 3, 6, and 12 months for the evaluation of optical density on the radiographs and the visual clinical interpretation of the remaining dentin as well as the evaluation using the radiographic subtraction method. The radiographic images from the different evaluation times will be scanned for the analysis of differences in density. For such, an specific program will be used.
Evaluation of time required for procedure | During the procedure.
  The time required for each procedure will be measured using a digital stopwatch (Kenko, Hong Kong) in minutes and seconds from the onset of treatment until the complete removal of the carious tissue. The time will be recorded on a specific chart for analysis.
Evaluation of need for local anesthesia during intervention | During the procedure.
  All interventions will be initiated without the prior administration of local anesthesia. The children will be told that anesthesia could be administered at any time during the intervention. The need for anesthesia, or not, will be recorded.
Changes in Clinical Evaluation | Immediately after treatment, 1 week, 1, 3, 6, and 12 months after treatment.
  The criteria used of the evaluation will be the retention of the restorative material in the cavity and the occurrence of secondary caries. Digital photographs of the restorations will also be taken and serve to complement the clinical and radiographic findings.
  0 = present; no defects;
  1. = present; small marginal defects measuring less than 0.5mm in depth; no need for repair;
  2. = present; small marginal defects measuring 0.5mm to 1mm in depth; need for repair;
  3. = present; large marginal defects measuring 1 or more mm in depth; need for repair;
  4. = absent; restoration nearly or completely lost; need for treatment;
  5. = absent; additional treatment having been performed for some reason;
  6. = tooth absent for any reason;
  7. = present; surface wear measuring less than 0.5mm in depth; no need for replacement;
  8. = present; surface wear greater than 0.5mm in depth; need for replacement;
  9. = impossible to diagnose.
Degree of pain/discomfort of children during procedure | During the procedure.
  A face scale with different expressions will be used and the child will be asked to point to the expression that most corresponds to his/her degree of pain/discomfort.
  Interpretation of face scale:
  1. No pain.
  2. Mild pain.
  3. Moderate pain.
  4. A little worse pain.
  5. Strong pain.
  6. Worst pain.

REFERENCES:
- [Derived] Martins LFB, de Sena LR, de Paula DM, Feitosa VP, Horliana ACRT, Fernandes KPS, Mesquita-Ferrari RA, Motta LJ, Goncalves MLL, Bussadori SK. Investigation on the effect of antimicrobial photodynamic therapy as an adjunct for management of deep caries lesions-study protocol for a randomized, parallel groups, controlled clinical trial. Trials. 2023 Mar 4;24(1):165. doi: 10.1186/s13063-023-07181-8. PMID 36870982